CLINICAL TRIAL: NCT01594606
Title: RCT of an Animal-Assisted Intervention With Adjudicated Youth
Brief Title: Randomized Control Trial of an Animal-Assisted Intervention With Adjudicated Youth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Annmarie Cano, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03HD070621 (NIH); R03HD070621 (NIH)
Record Dates: First submitted 2012-05-04; First posted 2012-05-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Conduct Disorder; Depression; Anxiety
Keywords: Animal-assisted intervention; adjudicated adolescents; empathy
MeSH Terms: conditions — Conduct Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Animal-assisted (Experimental): This group receives the dog training program in which they will be teaching a dog basic obedience skills.
  Interventions: Behavioral: Animal-assisted intervention
- Dog Walking (Active Comparator): This group will walk a different dog each week but will not engage in dog training.
  Interventions: Behavioral: Animal-assisted intervention

INTERVENTIONS:
Behavioral: Animal-assisted intervention — The experimental group will receive 10 weeks of classroom training and hands-on experience working with dogs to teach them basic obedience skills. Each participant will work with the same dog each week. The active control group will receive 10 weeks of classroom training and will walk a different dog each week but will not teach obedience skills to the dogs.

SUMMARY:
The project involves testing the efficacy of an animal-assisted intervention (AAI). The AAI consists of a 10-week program in which adjudicated adolescents train shelter dogs and will be compared to a dog walking control group matched for educational content and dog contact time. The investigators expect that the AAI will result in improved empathy skills and that dog attachment will explain these findings. The investigators also explore the extent to which the AAI will improve internalizing and externalizing symptoms in these adolescents.

DETAILED DESCRIPTION:
Adjudicated adolescents (i.e., teens who have committed criminal offenses and are incarcerated in juvenile detention centers) have deficits in emotion regulation, including empathy skills, and are at risk for a host of poor outcomes including repeat offenses, internalizing symptoms (e.g., depression, anxiety), externalizing symptoms (e.g., lying, truancy, fighting). Many of these problems stem from a lack of secure attachment to parents and peers. There is a need for novel and innovative programs to help these teens develop more secure attachments and better empathy skills to prevent poor outcomes. One type of intervention is animal-assisted interventions such as dog training programs. These programs appear to build empathy skills in at-risk youth, which may translate into better peer relations, less psychological distress, and less recidivism. The goal of this study is to test an existing animal-assisted intervention program that is already being used in juvenile detention centers to determine whether it is efficacious in improving adjudicated adolescents' empathy skills and psychological symptoms through building a secure attachment to the training dog.

ELIGIBILITY:
Inclusion Criteria:

* must be a resident of participating juvenile justice center in Michigan

Exclusion Criteria:

* none

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Internalizing and Externalizing Symptoms as measured by the Achenbach Child Behavior Checklist-Teacher Report and Youth Self Report forms | baseline and 10 weeks
  The Achenbach Child Behavior Checklist is a standardized measure of child behavior problems that assesses observers' and children's reports of the children's anxiety and depression (internalizing) and acting out (externalizing) behaviors.

SECONDARY OUTCOMES:
Change in empathy toward other people | baseline and 10 weeks
  An observational measure was created for the purposes of this study in which a trained confederate acts as a potential student for the animal-assisted intervention. The confederate will express anxiety about the program and the participants' responses will be coded by trained raters for empathic content.

CONTACTS AND LOCATIONS:
Overall Officials: Annmarie Cano, PhD, Principal Investigator — Wayne State University
Locations (1):
- Macomb County Juvenile Justice Center, Mount Clemens, Michigan, United States